CLINICAL TRIAL: NCT01772017
Title: A Multi Center, Open Label Study to Evaluate a Tongue Advancement Retainer Device in the Treatment of Subjects With Obstructive Sleep Apnea and Snoring (OPEN Trial)
Brief Title: A Trial to Evaluate a Device for the Treatment of OSA and Snoring
Acronym: OPEN
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decided to discontinue study for business reasons.
Sponsor: Sleepy, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OPEN-002
Record Dates: First submitted 2012-10-30; First posted 2013-01-21 (Estimated); Last update posted 2015-11-24 (Estimated); Status verified 2015-11

CONDITIONS: Obstructive Sleep Apnea; Snoring
Keywords: Obstructive Sleep Apnea; OSA; Snoring; Tongue Advancement Retainer Device
MeSH Terms: conditions — Sleep Apnea, Obstructive; Snoring

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Device Treatment (Experimental): Tongue Advancement Retainer Device
  Interventions: Device: Tongue Advancement Retainer Device

INTERVENTIONS:
Device: Tongue Advancement Retainer Device — Tongue Advancement Retainer Device
  Other Names: Sleepy Tongue Advancement Retainer Device

SUMMARY:
To evaluate the safety and efficacy of the Tongue Advancement Retainer Device in treating subjects with Obstructive Sleep Apnea (OSA) and snoring.

DETAILED DESCRIPTION:
The Tongue Advancement Retainer Device is a device that was developed to treat subjects with OSA and snoring. The purpose of this study is to evaluate initial safety and effectiveness of this device in treating one or both conditions.

ELIGIBILITY:
Inclusion Criteria:

* • Aged 18-65

  * AHI greater than or equal to 10 but less than or equal to 60 (<10 AHI <60/hr)
  * Complete set of lower anterior incisors with no evidence of periodontal disease or mobility and the ability to floss between teeth

Additionally subjects will in the screening phase must:

* Tolerate the device when being fitted
* Used the device for >4 hours on at least two consecutive nights during the screening period.
* Be able to reliably demonstrate proper installation of the device after fitting.
* Be willing to trial the device for a 4 week period

Exclusion Criteria:

* • Central sleep apnea events >10% of the total events

  * Evidence of Cheyne stokes breathing
  * Currently on treatment for OSA or OSA treatment discontinued less than 3 months prior.
  * Currently on regular treatment with prescription hypnosedatives or prescription stimulants
  * Very severe OSA, defined as AHI>60/hour and/or minimum oxygen saturation <75%
  * Need for immediate initiation of treatment as assessed by physician (e.g. Excessive sleepiness posing driving risk)
  * Previous surgery to treat OSA (other than nasal surgery)
  * Evidence of periodontal disease or tooth mobility
  * Severe nasal obstruction or enlarged tonsils based on clinical assessment
  * Unstable cardiovascular disease (untreated hypertension acceptable).
  * Inability to tolerate oral device due to oral condition or claustrophobia as determined by the study investigator
  * Pregnant/Breast Feeding
  * Any known factor or disease that might interfere with treatment compliance, study conduct or interpretation of the results such as co-existent other sleep disorder, psychiatric disease, history of non compliance to medical regimens, or unwillingness to comply with study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-10; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint - The safety of the device will be measured through recorded observations of adverse events. | Approximately 6 weeks
  Safety endpoint will be measured throughout the duration of the study.

SECONDARY OUTCOMES:
Primary Efficacy Endpoint - Change in the overall Apnea Hypopnea Index (AHI) from the PSG at baseline and end of treatment phase. | Approximately 6 weeks
  Efficacy Endpoint will be measured at baseline and at end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Brian Weeks, MD, Principal Investigator — Senta Clinic
Locations (3):
- United States (2):
  - Senta Clinic, San Diego, California
  - Visalia Medical Clinic, Visalia, California
- Royal North Shore Hospital, St Leonards, New South Wales, Australia